CLINICAL TRIAL: NCT05872269
Title: A Phase 4, Non-randomized, Multicentre, Open-label, Single-arm Study to Evaluate the Safety and Efficacy of Saroglitazar 4 mg in Patients With Non Alcoholic Fatty Liver Disease (NAFLD) With Comorbidities (Either Obesity, Type 2 Diabetes Mellitus, Dyslipidemia or Metabolic Syndrome)
Brief Title: A Study to Evaluate the Safety and Effectiveness of Saroglitazar 4 mg in Patients With NAFLD With Comorbidities
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARO.21.003
Record Dates: First submitted 2023-05-13; First posted 2023-05-24 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: NAFLD; Obesity; Type 2 Diabetes; Dyslipidemias; Metabolic Syndrome
Keywords: Real World Evidence Study
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Diabetes Mellitus, Type 2; Dyslipidemias; Metabolic Syndrome | interventions — saroglitazar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Saroglitazar 4 mg tablets (Experimental): Oral (once daily ) during 364 days/52 weeks of treatment period.
  Interventions: Drug: Saroglitazar

INTERVENTIONS:
Drug: Saroglitazar — 4 Mg Oral Tablet

SUMMARY:
A Phase 4, non-randomized, multicentre, open-label, single-arm study to evaluate the safety and efficacy of Saroglitazar 4 mg in patients with non-alcoholic fatty liver disease (NAFLD) with comorbidities (either obesity, type 2 diabetes mellitus, dyslipidemia or metabolic syndrome).

DETAILED DESCRIPTION:
The study is being planned to evaluate long term safety and efficacy of Saroglitazar 4 mg in patients with non-alcoholic fatty liver disease (NAFLD).

Total 1500 male and female patients with NAFLD with comorbidities (either obesity, type 2 diabetes mellitus, dyslipidemia or metabolic syndrome).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥18 years
2. Patients who have been prescribed Saroglitazar for NAFLD will be included in this Phase 4 study (patients who use Saroglitazar for the first time)
3. Patients able to and willing to provide written informed consent and comply with the requirements of the study protocol

   .
4. Patients with a prior documented diagnosis of NAFLD based on the AASLD criteria. NAFLD is defined either by previous histology or clinical imaging in individuals who consume little or no alcohol and do not have a cause for secondary hepatic steatosis or another cause of chronic liver disease. In addition, patients must have one of the following criteria to indicate ongoing NAFLD at screening:

   1. Liver stiffness through transient elastography, an LSM ≥8 kPa OR
   2. Serum ALT ≥45 U/L

Exclusion Criteria:

1. Consumption of alcohol for at least 90 consecutive days in last one year: >2 units of alcohol per day (>14 units per week) for males and >1 unit of alcohol per day (>7 units per week) for females. Note: 1 unit = 360 mL of beer, or 120 mL of wine, or 30 mL of spirits/hard liquor
2. History of other chronic liver disease (Viral hepatitis B or C, autoimmune hepatitis, cholestatic and metabolic liver diseases) and haemochromatosis.
3. Patient has known documented cirrhosis, either based on clinical criteria or liver histology or imaging.
4. Contraindications to Saroglitazar or any disease conditions affecting the ability to evaluate the effects of Saroglitazar.
5. History or other evidences of severe illness or any other conditions that would make patient, in the opinion of the investigator, unsuitable for the study.
6. Any previous history of ascites, hepatic encephalopathy, oesophageal varices or admission/emergency department visit for hepatic decompensation.
7. Women of child bearing potential: inability or unwillingness to practice contraception for the duration of the study.
8. Pregnant or breast feeding females

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Change in liver stiffness | Baseline to Week 52
  liver stiffness measurement performed by transient elastography
Frequency and severity of treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (TESAEs) | Baseline to Week 52

SECONDARY OUTCOMES:
Change in TG, HDL-C, LDL-C and non HDL-C levels | Baseline to Week 24 and Week 52
Change in serum ALT value | Baseline to Week 24 and Week 52
Change in serum AST value | Baseline to Week 24 and Week 52
Change in serum ALP value | Baseline to Week 24 and Week 52
Change in body weight | Baseline to Week 24 and Week 52
Change in BMI | Baseline to Week 24 and Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Deven Parmar, MD,FCP, Study Chair — Zydus Therapeutics Inc.
Locations (19):
- India (19):
  - Gastroplus Digestive Disease Centre, Ahmedabad
  - Mission GastroHospital, Ahmedabad
  - Artemis Hospital, Gūrgaon
  - Medanta- TheMedicity, Gūrgaon
  - Malla ReddyNarayanaMultispecialtyHospital, Hyderabad
  - Osmania GeneralHospital, Hyderabad
  - Yashoda Hospitals, Hyderabad
  - CARE CHL -Hospitals (Unit ofConvenient HospitalLtd., Indore
  - S R Kalla MemorialGastro and GenralHospital, Jaipur
  - AIIMS, Khorda
  - Medanta Hospital, Lucknow
  - Dayanand MedicalCollege & Hospital, Ludhiāna
  - Neurociti Hospital, Ludhiāna
  - TNMC & BYL NairCh. Hospital, Mumbai
  - Shree Siddhivinayak Maternity & Nursing Home, Nashik
  - Sir GangaramHospital, New Delhi
  - Alchemist Hospital, Panchkula
  - Fortis Hospital, Rupnagar
  - BAPS Pramukh Swami Hospital, Sūrat

IPD SHARING:
Plan to Share IPD: No